CLINICAL TRIAL: NCT01862536
Title: Tadalafil for Pulmonary Hypertension Associated With Chronic Lung Disease
Brief Title: Tadalafil for Pulmonary Hypertension Due to Chronic Lung Disease
Acronym: TADA-PHILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLIN-008-12F
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Results first posted 2021-03-09 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-02

CONDITIONS: Pulmonary Hypertension; Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Randomized trial; COPD; tadalafil; Phosphodiesterase inhibitor; Pulmonary hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Disease, Chronic Obstructive | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet
  Interventions: Drug: placebo
- Tadalafil (Experimental): Daily use of tadalafil (study drug) at 40 mg orally.
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — Daily use of study drug to treat pulmonary hypertension.
  Other Names: Cialis
  Arms: Tadalafil
Drug: placebo — Daily use in double blind study.
  Arms: Placebo

SUMMARY:
The functional, social, and economic burden of chronic obstructive lung disease (COPD) on the healthcare system is extraordinary. COPD is the fourth leading cause of death in the United States, and some estimates attribute up to $33.2 billion in health care costs to COPD-associated morbidity and mortality annually. The burden of COPD to the VA Healthcare system parallels these findings. According to the VA HSR&D Health Economics Resource Center, COPD ranks 5th among the 40 most common chronic clinical conditions in the U.S. Veteran patient population, is responsible for >14,000 VA hospital admission annually, and increases by $1,051/patient the total annual health care cost burden on the VA Healthcare system. Importantly, COPD is associated with frequent emergency room visitation and/or hospitalization patients. Pulmonary hypertension is a common co-morbid condition that worsen morbidity and mortality in patients with COPD. This study will examine the potential for tadalafil, a phosphodiesterase type-5 (PDE-5) inhibitor to improve functional status by decreasing pulmonary hypertension. Results from this study are expected to define the potential use of PDE-5 inhibitors in COPD-induced pulmonary hypertension. If successful, this treatment option may improve quality of life and outcomes for the large number of Veterans afflicted with PH due to COPD.

DETAILED DESCRIPTION:
Project Summary/Abstract This VA CSR&D Merit Review Award for a Clinical Trial proposal describes a 5-year program to support a prospective, placebo-controlled, randomized clinical trial (RCT) evaluating the effect of phosphodiesterase type-5 (PDE-5) inhibition with tadalafil at 40 mg daily over 12 months on exercise capacity in patients with at least moderate pulmonary hypertension (PH) PH (mean pulmonary artery pressure (mPAP) > 25 mm Hg, pulmonary vascular resistance (PVR)>3.0 Woods units, pulmonary capillary wedge pressure (PCWP) <18 mm Hg) due to chronic obstructive pulmonary disease (COPD) GOLD stage II or higher, FEV1FVC <70). PDE-5 inhibitors are recommended for World Health Organization (WHO) Category 1 PH but there is no evidence based recommendation supporting the use of these inhibitors in COPD-induced PH (WHO Category 3). In order to ensure maximum patient enrollment and to increase the clinical and demographic diversity of patients included in this study, the proposed research will be conducted at four VA sites: Boston VA Healthcare System, Providence VA Medical Center, the Greater Los Angeles VA Healthcare System , Atlanta VA and Denver VA. The research team includes senior investigators with extensive experience in the clinical management of patients with COPD and PH. The principal investigators (PI) for this study is Dr. Ronald H. Goldstein (Chief, Pulmonary Medicine at the Boston Healthcare System) and Dr Sharon Rounds (Chief, Medical Service, Providence VA). Dr Shelley Shapiro will serve as site PI at the Greater Los Angeles VA Healthcare System.

Within the Veteran population, COPD ranks among the most common chronic diseases and inflicts a substantial clinical and economic burden on the VA Healthcare System. Importantly, the vast majority of COPD-associated mortality and morbidity, including hospital admissions, is derived from a relatively select subpopulation of patients. There is emerging evidence to suggest that clinically evident PH is a key determinate of risk in COPD for exacerbations and progression of disease. The investigators found that moderate or severe PH is associated with significantly increased rates of COPD-related hospital readmission as compared to similar Veterans with COPD and only mild PH. Moreover, this trend was not influenced by differences in conventional measures of COPD disease severity (i.e., forced expiratory volume in 1 second [FEV1]) and was irrespective of supplemental oxygen status. These observations are in support of previously established clinical observations from others demonstrating that traditional COPD therapies, including supplemental oxygen, are ineffective at modulating sustained improvements to cardiopulmonary hemodynamics in patients with COPD and PH. It is established in specific forms of PH in which hypoxia is not the central mediator of disease progression that restoration of NO--dependent signaling in pulmonary vascular tissue is effective at attenuating pulmonary vascular remodeling to improve cardiopulmonary hemodynamics, exercise tolerance, and quality of life. The extent to which therapies that preserve NO--dependent signaling in pulmonary vascular tissue are effective in PH due to chronic lung disease, however, is not known.

Under physiological conditions, the enzyme phosphodiesterase type-5 (PDE-5) functions to maintain pulmonary vascular tone by degrading cGMP a key signaling intermediary involved in NO--dependent signaling. However, in PH due to lung disease, pulmonary vascular levels of NO- are diminished while PDE-5 levels are increased. This raises the possibility that PDE-5 inhibition is a potential strategy by which to increase NO- bioavailability and attenuate PH in patients with COPD, and sets the framework for the central hypothesis of the current proposal is that pharmacological inhibition of PDE-5 will improve functional capacity as assessed by 6 minute walk test in patients with COPD-induced moderate to severe PH. The secondary outcome measures will assess whether this change in functional status is accompanied by an improvement in maximal oxygen uptake during cardiopulmonary testing (VO2) and changes in vascular remodeling as assessed by cardiopulmonary hemodynamics. To test this hypothesis, a RCT will be conducted using tadalafil (40 mg orally daily) or placebo. The primary outcome measurements will be the six minute walk test. The secondary outcome measures will be functional assessment using peak volume of oxygen consumption (VO2) and the hemodynamic measures of PVR and mPAP. Additional information will be obtained related to the non-invasive assessment of pulmonary artery systolic pressure and right ventricular (RV) function including tricuspid annular plane systolic excursion, pulmonary artery acceleration time, and changes to the pulmonary outflow tract Doppler envelope, dyspnea, health related quality of life assessed by validated standardized questionnaires and the frequency of COPD exacerbations after 12 months. Results from this study are expected to define the potential use of PDE-5 inhibitors in COPD-induced PH. If successful, this treatment option may improve quality of life and outcomes for the large number of Veterans afflicted with PH due to COPD.

ELIGIBILITY:
Inclusion Criteria:

* Male and female U.S. Veteran patients 40-85 years old, with Gold Stage II COPD by pulmonary function testing (FEV1/FVC <0.70; performed within 6 months of recruitment.
* Eligible subjects must have PH documented on transthoracic echocardiogram within 6 months of baseline visit demonstrating an RV systolic pressure >40mmHg. To confirm the presence of PH, a right-heart catheterization will be performed, with subjects randomized to treatment only if catheterization shows a:

  * mPAP >25 mm Hg
  * PVR >2.5 Wood units
  * pulmonary artery capillary wedge pressure 18 mm Hg or less at rest
* PH belonging to the following subgroup of the updated Dana Point Clinical Classification:

  * Group 3 (PH associated with lung disease and/or hypoxemia) specifically, Group 3.1 (chronic obstructive pulmonary disease [COPD]) as the major criteria. Patients may also have minor clinical features associated with 3.2 (Interstitial disease) (such as mild fibrosis on high resolution chest CT, but total lung capacity>80% predicted) and 3.3 (sleep disordered breathing) (AHI <15 or 20/hour).
* 6-minute walk distance between 50-450 meters at screening visit.

Exclusion Criteria:

* PH belonging to the following subgroups of the updated Dana Point Clinical Classification:

Group 1

* Idiopathic
* heritable
* drug or toxin-induced
* Associated Pulmonary Arterial Hypertension (APAH) with:

  * connective tissue disease
  * congenital heart disease
  * or HIV

Group 2

* left atrial hypertension

Group 4

* chronic thromboembolic PH
* or other forms of PH not associated with primary lung disease

Also

* Patients with a history of systemic hypotension in the ambulatory setting (reproducible measurements of systolic blood pressure <89 mmHg) on chart review.
* Patients with moderate or severe hepatic impairment (Child-Pugh B and C)
* Patients with severe renal insufficiency (GFR <30 ml/min/1.73 m2)
* Severe aortic stenosis (aortic valve area <1.0 cm2)
* Patients with any acute or chronic impairment:

  * (other than dyspnea), limiting the ability to comply with the study requirements, including the 6-minute walk test and right heart catheterization.
* Patients with a recent stroke
* Patients with untreated hypoxemia (SaO2 <92%) at rest
* Patients with untreated moderate or severe obstructive sleep apnea (AHI>15)
* Patients with any coagulopathy
* Patients requiring nitrate therapy for any clinical indication
* Patients with an active prescription for pulmonary vasodilator medication other than oxygen
* Patients with a history of nonarteritic anterior ischemic optic neuropathy
* Contraindication to tadalafil use including allergy to:

  * any PDE-5 inhibitor
  * anatomical deformations of the penis
  * sickle cell anemia
  * multiple myeloma
  * leukemia
  * bleeding disorders
  * active peptic ulcer disease
  * retinitis pigmentosa or other retinal disorders.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H Goldstein, MD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (5):
- United States (5):
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, CO, Denver, Colorado
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
The PI will create de-identified, study-specific datasets. The PI will replace social security and medical station numbers with study-specific numbers.
  * A local privacy officer will certify that a dataset contains no PHI, PII, or VA Sensitive Information prior to release outside VA.
  * Final data sets will be maintained locally on a secure server or comparable data storage appliance inside the VA network until enterprise-level resources become available for long-term storage and access.
Time Frame: - Datasets meeting VA standards for disclosure to the public will be made available within 1 year of publication.
Access Criteria: Investigators requesting a copy of a dataset will sign a Letter of Agreement or a Data Use Agreement. The recipient will not attempt to identify any individual whose data are in the dataset. A local privacy officer will certify that a dataset contains no PHI, PII, or VA Sensitive Information prior to release outside VA.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The discrepancy between the enrollment number (44) and number in the participant flow module (36) was due to participant drop out. Of the 44 consented, 3 declined to participate, 3 did not complete the test dose trial, 1 had a medication conflict and 1 died prior to trial initiation.
Period: Overall Study
Arm/Group | Placebo | Tadalafil
Started | 13 | 23
Completed | 10 | 16
Not Completed | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tadalafil | Total
Number analyzed (Participants) | 13 | 23 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 8 | 14
  >=65 years | 7 | 15 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 13 | 23 | 36
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 23 | 36
6 Minute Walk Test [Median (Inter-Quartile Range); unit: Meters walked in 6 minutes] | 243.50 [182.90 to 317.00] | 249.35 [189.6 to 319.4] | 246.425 [186.85 to 318.20]

OUTCOME MEASURES:

1. Primary Outcome: Change in 6 Minute Walk Test
Description: Change from baseline in distance walked in 6 minutes.
Time Frame: The change in distance walked when assessed at 3 months following trial initiation as compared to baseline, similarly at 6 months compared to baseline, at 9 months compared to baseline and at 12 months compared to baseline.
Population: .The Overall Number of Participants Analyzed differs with the number in the Participant Flow because of subject drop out over the study period
Measure: Median (Inter-Quartile Range); unit: Meters walked in 6 minutes
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 13 | 19
Meters walked in 6 minutes
  Change in 6 MWT from baseline to 3 months | 7.00 [-2.70 to 28.00] | 16.60 [-15.20 to 48.19]
  Change in 6 MWT from baseline to 6 months: number analyzed (Participants) | 11 | 19
  Change in 6 MWT from baseline to 6 months | 16.00 [-12.00 to 42.00] | 4.90 [-23.40 to 45.12]
  Change in 6 MWT from baseline to 9 months: number analyzed (Participants) | 9 | 16
  Change in 6 MWT from baseline to 9 months | -18.00 [-61.00 to 32.00] | 8.93 [-24.45 to 54.10]
  Change in 6 MWT from baseline to 12 months: number analyzed (Participants) | 9 | 15
  Change in 6 MWT from baseline to 12 months | 21.00 [-9.00 to 40.00] | 16.76 [-1.70 to 49.30]

2. Secondary Outcome: Maximum VO2
Description: Measure of aerobic fitness on exercise assessed by cardiopulmonary exercise test.
Time Frame: 12 months
Population: The Overall Number of Participants Analyzed differs with the number in the Participant Flow because of subject drop out and patients who required supplemental oxygen did not have a cardiopulmonary exercise test performed.
Measure: Median (Inter-Quartile Range); unit: mL/kg/min
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 0 | 3
mL/kg/min |  | 13.6 [10.3 to 15.2]

3. Secondary Outcome: Pulmonary Vascular Resistance
Description: Pulmonary vascular resistance assessed on right heart catheterization is a hemodynamic measurement of pulmonary vascular remodeling.
Time Frame: 6 months
Population: The Overall Number of Participants Analyzed differs with the number in the Participant Flow because these participants refused to have a RHC procedure at the 12 month timepoint and therefore the PVR data was not available for analysis.
Measure: Median (Inter-Quartile Range); unit: mmHg
Groups:
- Tadalafil: Daily use of tadalafil (study drug) at 40 mg. orally
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 12 | 17
mmHg | 4.26 [2.93 to 5.83] | 2.69 [1.87 to 3.70]

4. Secondary Outcome: Mean Pulmonary Artery Pressure
Description: Mean pulmonary artery pressure assessed by right heart catheterization is a hemodynamic measurement of pulmonary hypertension severity.
Time Frame: 6 months
Population: The Overall Number of Participants Analyzed differs with the number in the Participant Flow because these participants refused to have a RHC procedure at the 12 month timepoint and therefore the mPAP data was not available for analysis.
Measure: Median (Inter-Quartile Range); unit: Wood units
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 12 | 17
Wood units | 33.00 [28.00 to 37.50] | 29.00 [25.00 to 38.00]

5. Secondary Outcome: Tricuspid Annular Plane Excursion (TAPSE)
Description: The tricuspid annular plane excursion is an echocardiographic measurement of right ventricular systolic dysfunction.
Time Frame: 12 months
Population: The Overall Number of Participants Analyzed differs with the number in the Participant Flow because these participants did not complete an ECHO procedure and therefore TAPSE data was not available for analysis.
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 8 | 14
mm | 2.08 [2.00 to 2.45] | 2.12 [1.70 to 2.30]

6. Secondary Outcome: St. George's Respiratory Questionnaire, Dyspnea and Health Related Quality of Life
Description: Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. There are 50 items, 2 parts, (3 components). Each item is accorded a weight determined by the degree of distress accorded to each symptom or state described.
  Scores range from 0-100, with higher scores indicating more limitations
Time Frame: 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 10 | 16
score on a scale | 49.34 [43.11 to 61.04] | 44.64 [36.26 to 55.68]

7. Secondary Outcome: N-type Brain Natriuretic Peptide (BNP) Concentration
Description: Plasma BNP concentration is a biochemical marker that correlates positively with pulmonary hypertension severity.
Time Frame: 12 months
Population: The Overall Number of Participants Analyzed differs with the number in the Participant Flow because these participants did not show up for the lab test and therefore the data was not available for analysis.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 9 | 14
pg/mL | 37.50 [26.00 to 365.2] | 47.81 [17.00 to 98.20]

8. Secondary Outcome: Resting Hypoxemia
Description: Changes to resting peripheral oxyhemoglobin saturation levels will be used to assess the safety of the study drug in patients with chronic lung diseases.
Time Frame: Early (4 hours and 3 days following treatment) and late (1, 3, 6, 9, 12 months following treatment)
Population: Measurements were not obtained
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Exercise-induced Hypoxemia
Description: Changes to peripheral oxyhemoglobin saturation levels on exercise will be used to assess the safety of the study drug in patients with chronic lung diseases.
Time Frame: 12 months
Population: Measurements were not obtained
Arm/Group | Placebo | Tadalafil
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo | Tadalafil
All-Cause Mortality (participants affected / at risk) | 1/13 | 5/23
Serious Adverse Events (participants affected / at risk) | 4/13 | 4/23
Other Adverse Events (participants affected / at risk) | 0/13 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | Tadalafil (N=23)
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) — not related to intervention
chest pain (Cardiac disorders) | 1 (1) | 2 (2) — not related to intervention
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — not related to intervention
hemoptysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — not related to intervention
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — not related to intervention
heartburn, dizziness, inability to swallow (General disorders) | 1 (1) | 4 (5) — not related to intervention
eye floaters (Eye disorders) | 0 (0) | 1 (1) — not related to intervention

LIMITATIONS AND CAVEATS:
This trial did not reach its enrollment goals. Enrollment was limited because of the unexpected frailty of patients with advanced COPD and evidence of elevated pulmonary artery pressure as assessed by cardiac echo. In addition we found that many potential candidates were found to have features of both group II and group III PH.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/36/NCT01862536/Prot_SAP_000.pdf